CLINICAL TRIAL: NCT07270939
Title: Optimizing Enteral Nutrition: A Comparative Study of 18-Hour, 20-Hour, and 24-Hour
Brief Title: Optimizing Enteral Nutrition Regimen for Critically Ill Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hamad Medical Corporation (Industry)
Responsible Party: Principal Investigator, Mr.Mutaz Ibrahim Omar Othman, Charge Nurse, Hamad Medical Corporation
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MRC-01-25-949
Record Dates: First submitted 2025-09-23; First posted 2025-12-08 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-11

CONDITIONS: Critical Illness; Enteral Nutrition; Ventilator Associated Pneumonia; Hyperglycemia; Feeding Intolerance
Keywords: Cyclic feeding; Feeding window; Critical care nutrition; Gastrointestinal tolerance; Nutritional adequacy
MeSH Terms: conditions — Critical Illness; Pneumonia, Ventilator-Associated; Hyperglycemia

STUDY DESIGN:
Intervention Model Description: Interventional Study Model: Parallel Assignment. Participants are randomized in a 1:1:1 ratio to one of three parallel groups (24-hour continuous feeding, 20-hour cycled feeding, 18-hour cycled feeding) and remain in their assigned group for the study duration.
Masking Description: Participants and clinical care teams will be aware of the assigned enteral feeding schedule. Outcome assessors and the statistician performing the final analysis will be blinded to group allocation where feasible.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 24-hour continuous feeding (control) (No Intervention): Feeding Schedule provides continuous enteral nutrition over 24 hours with no fasting window. This standard care in many ICUs serves as the baseline for comparison with two experimental cycled feeding regimens. The feeding rate is designed to evenly deliver the total daily caloric goal across the entire period.
- 20-hour cycled feeding (intervention) (Active Comparator): Feeding Schedule consists of enteral nutrition delivered over 20 hours, with a structured 4-hour fasting window each day. This approach aims to balance metabolic and gastrointestinal benefits while ensuring adequate daily caloric intake. Consequently, the feeding rate is increased to meet the total caloric goal within the shorter feeding period.
  Interventions: Behavioral: 20-Hour Cycled Enteral Nutrition with a 4-Hour Fasting Window
- 18-hour cycled feeding (intervention) (Active Comparator): Feeding Schedule involves enteral nutrition over an 18-hour period while incorporating a 6-hour fasting window in each 24-hour cycle. This structure is designed to test a more intense intermittent fasting regimen, aiming to enhance physiological benefits by better aligning with circadian rhythms. The expectations include improved metabolic control, enhanced gastrointestinal motility, and reduced infection rates, with careful monitoring for reduced caloric intake risk. Consequently, the feeding rate is increased to meet daily caloric goals within the 18-hour timeframe, resulting in the most intensive feeding schedule among the three examined arms.
  Interventions: Behavioral: 18-Hour Cycled Enteral Nutrition with a 6-Hour Fasting Window

INTERVENTIONS:
Behavioral: 20-Hour Cycled Enteral Nutrition with a 4-Hour Fasting Window — 20-Hour Cycled Enteral Nutrition with a 4-Hour Fasting Window (Intervention 1) Objective: To evaluate the physiological benefits of a structured daily fasting period while maintaining a conservative approach to caloric delivery.
  Other Names: Group Intervention 1
  Arms: 20-hour cycled feeding (intervention)
Behavioral: 18-Hour Cycled Enteral Nutrition with a 6-Hour Fasting Window — Feeding Schedule involves enteral nutrition over an 18-hour period while incorporating a 6-hour fasting window in each 24-hour cycle. This structure is designed to test a more intense intermittent fasting regimen, aiming to enhance physiological benefits by better aligning with circadian rhythms. The expectations include improved metabolic control, enhanced gastrointestinal motility, and reduced infection rates, with careful monitoring for reduced caloric intake risk. Consequently, the feeding rate is increased to meet daily caloric goals within the 18-hour timeframe, resulting in the most intensive feeding schedule among the three examined arms.
  Other Names: Group Intervention 2
  Arms: 18-hour cycled feeding (intervention)

SUMMARY:
Clinical Trial The goal of this clinical trial is to learn whether different enteral feeding cycles (18-hour, 20-hour, or standard 24-hour continuous feeding) improve outcomes for critically ill ICU patients who need tube feeding. It will also look at tolerance, nutrition delivery, and safety.

The main questions it aims to answer are:

Do shorter feeding cycles (with fasting windows) reduce ICU length of stay?

Do they lower the risk of infections like ventilator-associated pneumonia?

How do they affect calorie delivery, blood sugar control, and gastrointestinal tolerance?

Researchers will compare:

Continuous 24-hour feeding (standard care)

20-hour feeding with a 4-hour fasting window

18-hour feeding with a 6-hour fasting window

Participants will:

Be critically ill adults in the ICU who require at least 7 days of enteral feeding

Be randomized to one of the three feeding schedules

Receive daily monitoring of calories, protein, blood sugar, and GI tolerance

Have outcomes measured, including ICU length of stay, infections, metabolic control, and feeding tolerance

DETAILED DESCRIPTION:
This randomized controlled trial will compare three enteral feeding regimens in critically ill ICU patients: standard 24-hour continuous feeding, 20-hour cycled feeding with a 4-hour fasting window, and 18-hour cycled feeding with a 6-hour fasting window. The rationale is that continuous feeding may impair metabolic regulation, increase insulin requirements, and contribute to gastrointestinal intolerance, while cycled feeding could better align with circadian rhythms, support metabolic balance, and reduce complications such as ventilator-associated pneumonia.

Approximately 150 adult patients who require enteral nutrition for at least seven days will be enrolled across Hamad Medical Corporation ICUs. Participants will be randomized in a 1:1:1 ratio using block randomization through REDCap to ensure allocation concealment. All groups will receive isocaloric enteral nutrition through nasogastric or orogastric tubes, with caloric and protein targets guided by indirect calorimetry or weight-based calculations.

Feeding plans will be initiated within 24 hours of ICU admission or stabilization. Patients assigned to the 18-hour and 20-hour arms will have structured fasting periods, while the control group will receive uninterrupted feeding. Daily assessments will capture nutritional delivery, gastrointestinal tolerance, and metabolic parameters, along with safety monitoring for adverse events. Data will be collected electronically via REDCap, de-identified, and audited regularly by the Clinical Trial Unit.

The study is designed to generate high-quality evidence on whether incorporating fasting windows into feeding schedules can optimize nutrition therapy, improve tolerance, reduce ICU stays, and minimize complications. Findings are expected to inform future ICU nutrition guidelines and contribute to the global discussion on intermittent versus continuous feeding practices.

ELIGIBILITY:
Inclusion Criteria

Participants must meet ALL of the following criteria to be eligible for the study:

1. Patients aged ≥ 18 years.
2. Patients expected to require enteral nutrition (EN) for ≥ 7 days.
3. Critically ill, mechanically ventilated patients in the ICU.
4. New patients initiating EN in the critical care unit.
5. Patients receiving EN via:

   * a nasogastric (NG) tube.
   * orogastric (OG) feeding tube.

Exclusion Criteria:

1. Patients with contraindications to enteral feeding or pre-existing gastrointestinal disorders, including:

   * Active GI bleeding.
   * Progressive GI disease.
   * Recent GI tract resection.
2. Indication for a special diet formula.
3. Need for a large volume of feeding (as determined by the clinical team).
4. Pre-existing hepatic failure.
5. Use of a nasojejunal tube, gastrostomy, or jejunostomy.
6. Pregnancy confirmed via β-hCG testing for women of childbearing potential.
7. Insulin-dependent diabetes mellitus.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-12-30 (Estimated); Primary Completion 2026-11-30 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
ICU Length of Stay (LOS) | From the date of randomization until the date of ICU discharge or transfer, assessed up to 90 days (or until hospital discharge if it occurs earlier).
  The total number of days a patient spends in the intensive care unit, calculated from the date of ICU admission to the date of discharge or transfer out of the ICU.

SECONDARY OUTCOMES:
Nosocomial Infection/Pneumonia Incidence | Assessed daily from Day 3 to Day 7.
  Infections acquired after 48 hours of hospital admission, specifically including Ventilator-Associated Pneumonia (VAP). Diagnosed based on CDC criteria (clinical signs, laboratory findings, and imaging).
Nutritional Adequacy | Calculated daily from Day 1 to Day 7
  The percentage of the prescribed daily caloric goal that is actually delivered to the patient.
Gastrointestinal Complications | Monitored daily from Day 1 to Day 7
  Adverse events related to feeding intolerance.
Gastric Emptying Index | Measured every 4 hours, daily from Day 1 to Day 7.
  A measure of gastrointestinal motility, indicated by delayed gastric emptying. Aspirate gastric contents via a nasogastric (NG) or orogastric (OG) tube at regular intervals (every 4 hours). gastric residual volume ≤ 500 mL, persistently high GRV (>500 mL) indicates delayed emptying.
Glycemic Control | Daily, from Day 1 to Day 7 of the intervention.
  The regulation of blood glucose levels during the enteral nutrition intervention period.Average daily blood glucose level (mmol/L or mg/dL), calculated from point-of-care testing performed throughout the day.
Insulin Requirement | Daily, from Day 1 to Day 7 of the intervention.
  The total daily exogenous insulin dose required to maintain blood glucose within target range.Total insulin dose administered per 24-hour period, measured in units.
Serum Creatinine level, measured in mg/dL (or µmol/L) | Measured daily from Day 1 to Day 7. The baseline value is recorded on Day 0.
  The change in serum creatinine concentration from baseline serves as a specific biomarker of glomerular filtration rate (GFR) and kidney function.
Blood Urea Nitrogen (BUN) level, measured in mg/dL (or mmol/L) | Measured daily from Day 1 to Day 7 of the intervention. The baseline value is recorded on Day 0.
  Change in blood urea nitrogen concentration from baseline, as a biomarker of nitrogenous waste accumulation influenced by renal function, protein catabolism, and hydration status.
Alanine Aminotransferase (ALT) level, measured in U/L | Measured daily from Day 1 to Day 7 of the intervention. The baseline value is recorded on Day 0.
  The change in serum alanine aminotransferase (ALT) concentration from baseline serves as a specific biomarker of hepatocellular injury.
Aspartate Aminotransferase (AST) level, measured in U/L | Measured daily from Day 1 to Day 7 of the intervention. The baseline value is recorded on Day 0.
  Change in serum aspartate aminotransferase (AST) concentration from baseline, as a biomarker of hepatic inflammation and injury.
Total Bilirubin level, measured in mg/dL (or µmol/L) | Measured daily from Day 1 to Day 7 of the intervention. The baseline value is recorded on Day 0.
  The change in serum total bilirubin concentration from baseline serves as a biomarker of hepatic excretory function and bile flow.

OTHER OUTCOMES:
Inflammatory Marker | Measured daily from Day 1 to Day 7.The baseline value is recorded on Day 0.
  Level of systemic inflammation by Inflammatory Markers (e.g., CRP)
Patient Tolerance | Measured daily from Day 1 to Day 7
  The ability to receive enteral nutrition without significant adverse effects.

IPD SHARING:
Plan to Share IPD: No
Data will be collected and de-identified, codes will be used to cover patient identifiers such as Name, HC no., DOB. Any link between code and identifier will be deleted at the end of the data collection and anonymized data will be kept for at least 5 years after study completion. Study participation is documented using a unique study ID (e.g., "EN-001") rather than patient names. Access to identifiers is restricted to the research team and audited by the clinical trial unit (CTU) in HMC. The data that will be collected for this study will remain confidential.